CLINICAL TRIAL: NCT06796985
Title: High-Density Surface Electromyography Guided Precision Botulinum Neurotoxin Injections to Manage Chronic Pelvic Floor Pain
Brief Title: Botox for Chronic Pelvic Pain
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Yingchun Zhang, Professor, University of Miami
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20240022; 7R01DK133800-03 (NIH)
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Pelvic Floor Disorders
MeSH Terms: conditions — Pelvic Floor Disorders | interventions — Botulinum Toxins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group A: Standard injection template followed by HD-sEMG guided injection (Experimental): Participants will be in this group for up to 15 months
  Interventions: Drug: Botulinum neurotoxin; Device: High Density Surface Electromyographic, precision botulinum neurotoxin injection guidance medical device
- Group B: HD-sEMG guided injection followed by standard injection template (Experimental): Participants will be in this group for up to 15 months
  Interventions: Drug: Botulinum neurotoxin; Device: High Density Surface Electromyographic, precision botulinum neurotoxin injection guidance medical device

INTERVENTIONS:
Drug: Botulinum neurotoxin — Botulinum neurotoxin will be injected into the pelvic floor muscles following either a standard template (standard injection arm), or guided using high-density surface EMG (guided arm). Participants will receive this drug twice throughout the duration of the study. Approximately 200 units of botulinum neurotoxin will be administered per injection.
Device: High Density Surface Electromyographic, precision botulinum neurotoxin injection guidance medical device — A personalized, precision botulinum neurotoxin injection guidance medical device, utilizing an intra-vaginal high-density surface EMG system to optimize the treatment outcomes in chronic pelvic pain (CPP) management. The device will be used five times during the study. Each use will last approximately ten minutes.

SUMMARY:
The purpose of this research study is to find out if precise, targeted injection of botulinum neurotoxin (commonly known as Botox) provides better relief of pelvic floor hypertonicity and pain than the standard method being used. The researchers want to better understand the effects (good and bad) of targeted botulinum neurotoxin injections in women with pelvic floor disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Females between 18 and 75 years of age
2. Clinical diagnosis of chronic pelvic pain
3. Complaints of pain, pressure, or discomfort in the bladder and/or pelvic area for the past 6 months or more, associated with lower urinary tract symptoms (such as frequency of urination), in the absence of other explanation of the symptoms (e.g., UTI) *
4. Myofascial pain diagnosed with palpable bands or nodules of contracted muscle fibers
5. Pelvic muscle tenderness by assessment of pelvic floor muscles on digital pelvic examination
6. No botulinum neurotoxin pelvic floor muscle injection treatment within 6 months prior to recruitment
7. Able to provide informed consent

Exclusion Criteria:

1. Males
2. Women < 18 and > 76 years of age
3. History of pelvic malignancy and sexual transmitted diseases that is currently not in remission
4. Bleeding disorder such as coagulopathy
5. Hypersensitivity to botulinum neurotoxin
6. Received botulinum neurotoxin pelvic floor muscle injection within 6 months prior to recruitment
7. History of neurological disorders, such as spinal cord injury, multiple sclerosis, amyotrophic lateral sclerosis or myasthenia gravis
8. Pregnancy, breast feeding or planning to get pregnant within one year after the last botulinum neurotoxin injection.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2027-03-22 (Estimated); Study Completion 2027-03-22 (Estimated)

PRIMARY OUTCOMES:
Hypertonic index of the pelvic muscles as measured by high-density surface-EMG (HD-sEMG) | 1 month post-injection
  The muscle hypertonicity Index measured by using HD-sEMG which is a ratio between the root mean square (RMS) of pelvic floor muscle EMG at rest and contraction.

SECONDARY OUTCOMES:
Change in Self-Report Pelvic Pain as measured by Global Response Assessment (GRA) | Baseline, 1 month post-injection
  Assessment is scored 0-6. Lower score indicates less pain while higher score indicates more pain.
Change in Self-Report Pelvic Symptoms as measured by Global Response Assessment (GRA) | Baseline, 1 month post-injection
  Assessment is scored 1-7. Lower score indicates worse symptoms while higher score indicates less symptoms.
Change in Self-Report Pelvic Pain as measured by the Female Genitourinary Index | Baseline, 1 month post-injection
  Sum score will be collected and scores range from 0-45. Lower score indicates less pain while higher score indicates more pain.

CONTACTS AND LOCATIONS:
Overall Officials: Yingchun Zhang, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No